CLINICAL TRIAL: NCT04834895
Title: Investigation of the Effectivenes of Digital Based Exercises in Patients With Neck Pain
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Marmara University (Other)
Responsible Party: Principal Investigator, Eda Tonga, Doctor of Philosopy, Marmara University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 09.2019.1056
Record Dates: First submitted 2021-02-21; First posted 2021-04-08 (Actual); Last update posted 2021-04-08 (Actual); Status verified 2021-04

CONDITIONS: Neck Pain
Keywords: Neck pain; exercise; digital health; mHealth; adherence
MeSH Terms: conditions — Neck Pain; Motor Activity

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- mhealth exercise group (Active Comparator): home exercise program is given to patients via mobile application
  Interventions: Other: mhealth exercise group
- brochure exercise group (Experimental): home exercise program is given to patients via brochure
  Interventions: Other: brochure exercise group

INTERVENTIONS:
Other: mhealth exercise group — Participants were asked to perform 18 exercises specially prepared for neck pain in the M.ü Neck Exercises application according to the number of repetitions specified in the application.Participants will be asked to do home exercises 3 days a week for 6 weeks
  Arms: mhealth exercise group
Other: brochure exercise group — Participants were asked to perform 18 exercises specially prepared for neck pain in the brochure according to the number of repetitions specified in the application.Participants will be asked to do home exercises 3 days a week for 6 weeks
  Arms: brochure exercise group

SUMMARY:
In study, the researchers examine the effectiveness of digital-based exercises in patients with chronic neck pain.The planned study has 2 main objectives:

* Increase exercise adherence with mhealth apps.
* To reduce pain and disability of patients with chronic neck pain.

DETAILED DESCRIPTION:
Neck pain is one of the most common musculoskeletal diseases after low back pain in the community. The incidence of neck pain was reported as %37,2. Neck pain can be caused by trauma, poor posture, degenerative diseases, tumors, muscle stress, wiplash injuries, cervical myelopathy, cervical ligamentous instability, fracture, vascular insufficiency or systemic diseases. Neck pain is classified as acute (less than six weeks), subacute (six to twelve weeks) or chronic (lasting more than twelve weeks). While neck pain is treated in physiotherapy clinics, it is also supported by home exercises during and after treatment.

It is emphasized that home exercise programs for neck pain are effective, but exercise adherence is an important factor. Nowadays, with the rapid development of mobile healthcare applications, digital based exercise applications have started to be used in physiotherapy and rehabilitation. Although it has been shown to be useful in studies examining the effectiveness of mHealth applications for different musculoskeletal problems, these studies are quite limited. Several studies have identified the beneficial effects of digital-based exercises, but no clear evidence of superiority over written or oral home exercise programs. In 2019, a mobile exercise application (Neck Exercise) for neck pain patients was developed as a thesis study at Marmara University Health Sciences Institute. The availability of this mobile application is shown on healthy people. However, its efficacy has not been studied in patients with chronic neck pain. This mobile app includes for the neck spinal stabilization , posture, breathing exercises and exercises for scapula circumference. Each exercise is explained with video. In addition, this application gives reminder signals at user-defined time intervals. Participants with chronic neck pain aged between 18-65 years will be included in the study and randomly divided into two groups. One group will be given home exercises via brochure to the other group via mobile application. Participants will be asked to do home exercises 3 days a week for 6 weeks. Pain, disability and exercise adherence of the participants will be evaluated. The Nordic Musculoskeletal Questionnaire, VAS, neck disability index and exercise adherence scale will be used in the evaluation. Our thesis will be the first study examining the effect of a mobile application developed for neck pain on adherence to home exercises. As a result of study, the researchers aim to save paper by prescribing home exercise programs via mobile application and to promote a platform where users can better understand the exercises.

ELIGIBILITY:
Inclusion Criteria:

* Neck pain that has been going on for at least 3 months
* Participant can use smart phone,
* No problem affecting reading and answering survey questions

Exclusion Criteria:

* Presence of visual and auditory problems that may prevent the use of the smartphone application
* Torticollis
* Vertigo
* Pregnancy
* Additional diseases such as vertebrobasilar insufficiency, heart failure, chronic heart disease and hypertension
* Dementia
* Inflammatory rheumatic disease
* Psychosis and neurological disease diagnosis
* Receiving another treatment or having surgery in 3 months
* Exposure to any neck trauma in the past 6 months
* A past or ongoing cancer history

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2021-02-01 (Actual); Primary Completion 2021-07-20 (Estimated); Study Completion 2021-07-30 (Estimated)

PRIMARY OUTCOMES:
Change from Visual Analog Scale (VAS) score at 6 Weeks | Baseline and Week 6
  VAS is the most commonly used method to assess pain intensity. The leftmost value in the 10 cm horizontal line used for VAS is scored between 0 cm (no pain) and the rightmost value is between 10 cm (unbearable pain) (Boonstra, Schiphorst Preuper et al. 2008). Measurements were recorded at the beginning and end of exercise training for both groups.
Change from Exercise Adherence Scale Points at 6 Weeks | Baseline and Week 6
  It consists of four yes / no questions.'Yes' answer is rated with 1 point, 'No' answer gets 0 point. Lesser scores indicate good exercise adherence.

SECONDARY OUTCOMES:
Change from Neck Pain and Disability Index Points at 6 Weeks | Baseline and Week 6
  Neck pain and disability balance consist of 20 items. Scoring of each item is done with a 10 cm visual analog scale and scored between 0 and 5 points. The Turkish version study of Biçer et al. Whose reliability and validity has been proven. It was made by (Biçer 2004). The items evaluate the severity of pain and the effect of pain on professional, recreational, social, daily life activities and their relationship with emotional factors. Thus, it measures the effects of neck pain on functionality, quality of life and disability. The total score is the sum of the points in each item and ranges from 0 to 100. The score evaluation was carried out as follows (Buko 2013).
  0-4: no problem 5-14: mild severity problem 15-24: moderate severity problem 25-34: severe problem 35 and above: very severe problem

OTHER OUTCOMES:
Change from The Nordic Musculoskeletal Questionnaire at 6 Weeks | Baseline and Week 6
  It is used to question musculoskeletal disorders. The Nordic Musculoskeletal Questionnaire, reliable information about the onset, prevalence and outcome of musculoskeletal pain in nine body areas (neck, shoulders, back, elbows, wrists / hands, waist, hips / thighs, knees, ankles / feet) Provider is a questionnaire that can be filled in by self or personal interview technique. The Nordic Musculoskeletal Questionnaire is a measure that can be used for musculoskeletal pain and related conditions in studies conducted in general and / or general communities. The Scandinavian musculoskeletal system query questions yes / no .

CONTACTS AND LOCATIONS:
Locations (1):
- Marmara University, Istanbul, Turkey (Türkiye)